CLINICAL TRIAL: NCT04529798
Title: A Monocentric Clinical Study Evaluating Clinical and Patient-reported Outcomes of Reverse Shoulder Arthroplasty With SMR Stemless
Brief Title: Clinical Study Evaluating Outcomes of Reverse Shoulder Arthroplasty With SMR Stemless
Acronym: SSPR
Status: Recruiting | Type: Observational
Sponsor: Arthro Medics AG (Other)
Responsible Party: Principal Investigator, Prof. Dr. med Claudio Rosso, Principal Investigator, Arthro Medics AG
Other Study IDs: S-35
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Rotator Cuff Tear Arthropathy; Osteo Arthritis Shoulders
Keywords: stemless reverse shoulder arthroplasty
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of this study are the assessment of the clinical, radiographical and patient-reported outcomes of SMR Stemless Reverse Shoulder Arthroplasty (LimaCorporate S.p.A.) used as standard of care over a period of at least 2 years of follow-up and the evaluation of the incidence of any complication.

DETAILED DESCRIPTION:
The focus of this study is the evaluation on clinical, patient-reported and radiographical outcomes of SMR Stemless Reverse Shoulder Arthroplasty. There is a retrospective and prospective study population.

The follow up time-points are (as of standard of care and not different for this study):

* Baseline
* 6 weeks postop
* 6 months postop
* 12 months postop
* 24 months postop

ELIGIBILITY:
Inclusion Criteria:

* rotator-cuff arthropathy, osteoarthritis
* approving written informed consent

Exclusion Criteria:

* Female patients who are pregnant, nursing, or planning a pregnancy.
* All adult patients with any of the SMR Stemless contraindication for use for the reverse configuration as reported in the current local Instruction for use.
* not consenting in participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There is a retrospective and prospective study population. All participants are older than 18 years old and approved the written informed consent. Additionally they are suffering from rotator-cuff arthropathy and/or osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11-22 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Subjective Shoulder Value score | 5 years
  Evaluation of the change of the Subjective Shoulder Value score from pre-operative to the last follow-up visit.

SECONDARY OUTCOMES:
ASES Shoulder Score | 5 years
  Evaluation of the change of the ASES shoulder score from pre-operative to the last follow-up visit.
Quick-Dash score | 5 years
  Evaluation of the change of the Quick-Dash score from pre-operative to the last follow-up visit.
VAS pain | 5 years
  Evaluation of the change of the VAS pain score from pre-operative to the last follow-up visit.
UCLA shoulder score | 5 years
  Evaluation of the change of the UCLA shoulder score from pre-operative to the last follow-up visit.
Loosening, implant stability, radiolucent lines | 1 year
  Radiographic evaluation of the implant stability as rate and progression of symptomatic radiolucent lines and loosening.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Rosso, Prof. Dr. med., Principal Investigator — Arthro Medics AG
Locations (1):
- Arthro Medics AG, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No